CLINICAL TRIAL: NCT00021164
Title: Immunization of HLA-A*0201 Patients With Metastatic Cancer Using a Peptide Epitope From the Telomerase Antigen
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068756; NCI-01-C-0176; NCI-4970; NCT00016640 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-04

CONDITIONS: Melanoma (Skin); Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV melanoma; recurrent melanoma; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; incomplete Freund's adjuvant

INTERVENTIONS:
Biological: aldesleukin
Biological: incomplete Freund's adjuvant
Biological: telomerase: 540-548 peptide vaccine

SUMMARY:
RATIONALE: Vaccines made from a peptide may make the body build an immune response and kill tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of vaccine therapy in treating patients who have metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether an immunologic response can be obtained in HLA*0201-expressing patients with metastatic cancer treated with telomerase: 540-548 peptide vaccine emulsified in Montanide ISA-51.
* Determine which vaccine strategy (frequency, schedule, and dosing) is best for future studies in these patients.
* Determine the toxicity of this treatment in these patients.
* Determine whether prior immunization with telomerase: 540-548 peptide vaccine results in increased clinical response to interleukin-2 in patients with melanoma.

OUTLINE: This is a randomized study. Patients are stratified according to disease (metastatic cutaneous melanoma vs other tumor types). Patients are randomized to one of three treatment arms.

* Arm I: Patients receive telomerase: 540-548 peptide vaccine emulsified in Montanide ISA-51 subcutaneously (SC) on day 1 of weeks 1-4 and 7-10. Patients also undergo leukapheresis over 3 hours at baseline and after each course of treatment.
* Arm II: Patients receive telomerase: 540-548 peptide vaccine emulsified in Montanide ISA-51 SC on day 1 of weeks 1, 4, 7, and 10. Patients also undergo leukapheresis over 3 hours at baseline, after the vaccine on week 4, and after each course of treatment.
* Arm III: Patients receive telomerase: 540-548 peptide vaccine emulsified in Montanide ISA-51 SC on days 1-4 of weeks 1, 4, 7, and 10. Patients undergo leukapheresis as in arm II.

Treatment in all arms repeats every 13 weeks for 4-6 courses in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 1 additional course of treatment after achieving CR.

Eligible melanoma patients with progressive disease on vaccine alone on any of the 3 arms may receive interleukin-2 (IL-2) combined with vaccine as in arm II. Beginning the day after each immunization, IL-2 is administered IV over 15 minutes every 8 hours over 4 days on weeks 1, 4, 7, and 10 for a maximum of 12 doses. Patients continuing to experience disease progression on combined vaccine and IL-2 therapy go off study after 2 courses of combined therapy.

Patients are followed at 3 weeks.

PROJECTED ACCRUAL: A total of 90-162 patients (30-54 per treatment arm; 45-81 per stratum) will be accrued for this study within less than 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Presenting with evaluable metastatic cancer

  * Refractory to standard treatment OR
  * Post-radiation for malignant glioma
* HLA-A*0201 expression

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 90,000/mm^3

Hepatic:

* Bilirubin no greater than 1.6 mg/dL
* AST/ALT less than 3 times normal
* Hepatitis B surface antigen negative

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No cardiac ischemia by stress thallium or comparable test*
* No prior myocardial infarction*
* No cardiac arrhythmias* NOTE: *Patients receiving interleukin-2 (IL-2) only

Pulmonary:

* No obstructive or restrictive pulmonary disease (patients receiving IL-2 only)

Immunologic:

* HIV negative
* No autoimmune disease or any other known immunodeficiency disease
* No active primary or secondary immunodeficiency

Other:

* No other active major medical illness*
* No active systemic infection
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception NOTE: *Patients receiving IL-2 only

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior telomerase: 540-548 peptide immunization

Chemotherapy:

* Recovered from prior chemotherapy

Endocrine therapy:

* No requirement for systemic steroid therapy

Radiotherapy:

* See Disease Characteristics
* Recovered from prior radiotherapy

Surgery:

* Not specified

Other:

* At least 3 weeks since prior systemic therapy for cancer

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-05; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States